CLINICAL TRIAL: NCT06902831
Title: Comparative Outcomes of Endoscopic and Open Carpal Tunnel Release with Neurotrophic Supplementation in Severe Carpal Tunnel Syndrome
Status: Completed | Type: Observational
Sponsor: University of Bari (Other)
Responsible Party: Principal Investigator, Rossella Elia, MD PhD, Prof. Rosella Elia, University of Bari
Other Study IDs: JHS-S-24-01434
Record Dates: First submitted 2025-02-25; First posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Carpal Tunnel Syndrome (CTS)
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Open Carpal Tunnel Release without Neurotrophic
  Interventions: Procedure: Open carpal tunnel release
- Endoscopic Carpal Tunnel Release without Neurotrophic
  Interventions: Procedure: Endoscopic Carpal Tunnel Release
- Open Carpal Tunnel Release with Neurotrophic
  Interventions: Procedure: Open carpal tunnel release; Drug: Neurotrophic supplementation
- Endoscopic Carpal Tunnel Release with Neurotrophic
  Interventions: Procedure: Endoscopic Carpal Tunnel Release; Drug: Neurotrophic supplementation

INTERVENTIONS:
Procedure: Endoscopic Carpal Tunnel Release — Release of carpal tunnel with endoscopic device
  Groups: Endoscopic Carpal Tunnel Release with Neurotrophic; Endoscopic Carpal Tunnel Release without Neurotrophic
Procedure: Open carpal tunnel release — Release of carpal tunnel with open tecnique
  Groups: Open Carpal Tunnel Release with Neurotrophic; Open Carpal Tunnel Release without Neurotrophic
Drug: Neurotrophic supplementation — Neurotrophic supplementation after surgery
  Groups: Endoscopic Carpal Tunnel Release with Neurotrophic; Open Carpal Tunnel Release with Neurotrophic

SUMMARY:
This study addresses the pressing clinical question of optimizing surgical and pharmacological interventions for severe Carpal Tunnel Syndrome (CTS), a prevalent and debilitating condition caused by median nerve compression. Previous research has established the efficacy of Open Carpal Tunnel Release (OCTR) and Endoscopic Carpal Tunnel Release (ECTR); however, the role of neurotrophic supplementation in enhancing surgical outcomes has yet to be fully elucidated. Using a prospective clinical approach involving 497 patients, we evaluated the comparative outcomes of ECTR and OCTR with or without neurotrophic supplementation. Key findings demonstrate that ECTR, particularly when combined with neurotrophic agents, facilitates faster recovery and greater improvements in Sensory Nerve Conduction Velocity (VCS) and Visual Analog Scale (VAS) scores, with reduced complication rates compared to OCTR

ELIGIBILITY:
Inclusion Criteria:

* clinically and electromyographically confirmed severe CTS (SCV < 35 m/s)
* experienced persistent symptoms unresponsive to conservative treatments for at least six months

Exclusion Criteria:

* mild or moderate CTS
* concomitant neuropathies
* previous carpal tunnel surgeries
* contraindications to neurotrophic supplementation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients diagnosed with severe Carpal Tunnel Syndrome from Policlinico of Bari
Sampling Method: Non-Probability Sample
Enrollment: 497 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
SCV evaluation | 12 months of follow-up
  SCV will be evaluated through electomyography after ECTR or OCTR with or without neurotrophic supplementation
VAS for pain evaluation | 12 months of follow-up
  VAS for pain will be evaluated through questionnarie after ECTR or OCTR with or without neurotrophic supplementation
VAS for funcionality evaluation | 12 months of follow-up
  VAS for functionality will be evaluated through questionnarie after ECTR or OCTR with or without neurotrophic supplementation

CONTACTS AND LOCATIONS:
Locations (1):
- Policlinico di Bari, Bari, Italy, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Desideri I, Francolini G, Becherini C, Terziani F, Delli Paoli C, Olmetto E, Loi M, Perna M, Meattini I, Scotti V, Greto D, Bonomo P, Sulprizio S, Livi L. Use of an alpha lipoic, methylsulfonylmethane and bromelain dietary supplement (Opera(R)) for chemotherapy-induced peripheral neuropathy management, a prospective study. Med Oncol. 2017 Mar;34(3):46. doi: 10.1007/s12032-017-0907-4. Epub 2017 Feb 15. PMID 28205185
- [Background] Nikbakht S, Vafaei MA, Ashraf A, Nasiri A, Nikpay-Hosseinabad N. Assessment of L-carnitine effectiveness on carpal tunnel syndrome. Curr J Neurol. 2022 Jul 6;21(3):162-169. doi: 10.18502/cjn.v21i3.11109. PMID 38011355
- [Background] Salehi B, Berkay Yilmaz Y, Antika G, Boyunegmez Tumer T, Fawzi Mahomoodally M, Lobine D, Akram M, Riaz M, Capanoglu E, Sharopov F, Martins N, Cho WC, Sharifi-Rad J. Insights on the Use of alpha-Lipoic Acid for Therapeutic Purposes. Biomolecules. 2019 Aug 9;9(8):356. doi: 10.3390/biom9080356. PMID 31405030
- [Background] Kim PT, Lee HJ, Kim TG, Jeon IH. Current approaches for carpal tunnel syndrome. Clin Orthop Surg. 2014 Sep;6(3):253-7. doi: 10.4055/cios.2014.6.3.253. Epub 2014 Aug 5. PMID 25177448
- [Background] Orhurhu V, Orman S, Peck J, Urits I, Orhurhu MS, Jones MR, Manchikanti L, Kaye AD, Odonkor C, Hirji S, Cornett EM, Imani F, Varrassi G, Viswanath O. Carpal Tunnel Release Surgery- A Systematic Review of Open and Endoscopic Approaches. Anesth Pain Med. 2020 Dec 26;10(6):e112291. doi: 10.5812/aapm.112291. eCollection 2020 Dec. PMID 34150584
- [Background] Zieske L, Ebersole GC, Davidge K, Fox I, Mackinnon SE. Revision carpal tunnel surgery: a 10-year review of intraoperative findings and outcomes. J Hand Surg Am. 2013 Aug;38(8):1530-9. doi: 10.1016/j.jhsa.2013.04.024. Epub 2013 Jun 25. PMID 23809470
- [Background] Sayegh ET, Strauch RJ. Open versus endoscopic carpal tunnel release: a meta-analysis of randomized controlled trials. Clin Orthop Relat Res. 2015 Mar;473(3):1120-32. doi: 10.1007/s11999-014-3835-z. Epub 2014 Aug 19. PMID 25135849
- [Background] Soltani AM, Allan BJ, Best MJ, Mir HS, Panthaki ZJ. A systematic review of the literature on the outcomes of treatment for recurrent and persistent carpal tunnel syndrome. Plast Reconstr Surg. 2013 Jul;132(1):114-121. doi: 10.1097/PRS.0b013e318290faba. PMID 23806914
- [Background] Means KR Jr, Dubin NH, Patel KM, Pletka JD. Long-term outcomes following single-portal endoscopic carpal tunnel release. Hand (N Y). 2014 Sep;9(3):384-8. doi: 10.1007/s11552-014-9614-1. PMID 25191172
- [Background] Atroshi I, Hofer M, Larsson GU, Ranstam J. Extended Follow-up of a Randomized Clinical Trial of Open vs Endoscopic Release Surgery for Carpal Tunnel Syndrome. JAMA. 2015 Oct 6;314(13):1399-401. doi: 10.1001/jama.2015.12208. No abstract available. PMID 26441187
- [Background] Marvulli R, Ianieri G, De Venuto G, Falcicchio M, Gallo GA, Mennuni C, Gallone MF, Fiore P, Ranieri M, Megna M. Electrophysiological and Clinical Improvement in Non-Invasive Treatment of Carpal Tunnel Syndrome. Endocr Metab Immune Disord Drug Targets. 2021;21(2):345-351. doi: 10.2174/1871530320666200728152953. PMID 32723265
- [Background] Stevens JC, Smith BE, Weaver AL, Bosch EP, Deen HG Jr, Wilkens JA. Symptoms of 100 patients with electromyographically verified carpal tunnel syndrome. Muscle Nerve. 1999 Oct;22(10):1448-56. doi: 10.1002/(sici)1097-4598(199910)22:103.0.co;2-y. PMID 10487914
- [Background] Nordstrom DL, DeStefano F, Vierkant RA, Layde PM. Incidence of diagnosed carpal tunnel syndrome in a general population. Epidemiology. 1998 May;9(3):342-5. PMID 9583428
- [Background] Mondelli M, Giannini F, Giacchi M. Carpal tunnel syndrome incidence in a general population. Neurology. 2002 Jan 22;58(2):289-94. doi: 10.1212/wnl.58.2.289. PMID 11805259
- [Background] Spahn G, Wollny J, Hartmann B, Schiele R, Hofmann GO. [Metaanalysis for the evaluation of risk factors for carpal tunnel syndrome (CTS) Part II. Occupational risk factors]. Z Orthop Unfall. 2012 Oct;150(5):516-24. doi: 10.1055/s-0032-1315346. Epub 2012 Oct 17. German. PMID 23076750